CLINICAL TRIAL: NCT02180958
Title: Evaluation of ONYX in ENDOVASCULAR Treatment of Cerebral AVMs. Prospective, Multi-center and Observational French Study
Brief Title: Evaluation of ONYX in ENDOVASCULAR Treatment of Cerebral AVMs
Acronym: cAVM
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-ONY-002
Record Dates: First submitted 2014-04-25; First posted 2014-07-03 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Arteriovenous Malformations
Keywords: cerebral arteriovenous malformations; cAVM; ONYX
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cerebral Arteriovenous Malformations: Adult patients requiring endovascular treatment of Cerebral Arteriovenous Malformations.

SUMMARY:
To assess safety and efficacy of ONYX treatment for cAVM:

DETAILED DESCRIPTION:
The main objective of this study is to assess the safety at 1 month after any embolization session and the efficacy at:

* 12 months post last embolization in case of treatment with embolization only
* 12 months after additional treatment with neurosurgery
* 36 months after additional treatment with radiosurgery

ELIGIBILITY:
Inclusion Criteria:

* The patient presents a cerebral AVM (not already treated) that can be treated by embolization with Onyx whether or not associated with a cyanoacrylate based adhesive,
* The patient is at least 6 years old.

Exclusion Criteria:

* During the treatment period for his/her cerebral AVM, the patient participates in a study assessing another medical device, another procedure or a drug.
* The patient and/or his/her legal representative (if applicable) refuses to give his/her consent to the collection and processing of data required by the centralized follow-up. For patients who refused collection of their personal data, only, the reason for non inclusion and date of implantation will be documented.
* Any condition that could prevent follow-up of the patient.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients from participating centres for whom a cerebral AVM (not already treated) has to be treated (whatever treatment method anticipated) and who do not object to the collection and transmission of data concerning them, will be included in the so-called "screened" population.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Device or procedure Adverse Events | 1 month
  Device or procedure related adverse events
Healing rate | 12 or 36 months
  No residual early venous return
  * 12 months after last embolization in case of complete treatment or stopping treatment;
  * 12 months after additional intervention in case of additional treatment required by neuro-surgery;
  * 36 months after additional intervention in case of additional treatment required by radio-surgery.

SECONDARY OUTCOMES:
Describe funtional independence | 1 and 12 months
  Describe mRS scores assessed by a certified physician

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Ricolfi, Prof. Dr., Principal Investigator — Centre Hospitalier Universitaire Dijon; Christophe Cognard, Prof. Dr., Principal Investigator — University Hospital, Toulouse; Laurent Spelle, Prof. Dr., Principal Investigator — Hôpital Bicêtre
Locations (17):
- France (17):
  - CHU Besançon, Besançon
  - Chu Pellegrin, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHI Dijon, Dijon
  - CHP Clairval, Marseille
  - Hôpital GUI DE CHAULLAC, Montpellier
  - CHU Nantes, Nantes
  - Fondation Ophtamoligique Rothschild, Paris
  - Groupe Hospitalier Pitier Salpetrière, Paris
  - Hôpital Beaujon, Paris
  - Hôpital Bicêtre, Paris
  - CHU Pontchaillou, Rennes
  - CHU Strasbourg, Strasbourg
  - HIA Sainte Anne, Toulon
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available